CLINICAL TRIAL: NCT02325518
Title: The Efficacy and Safety of Brinzolamide 1%/Timolol 0.5% Fixed Combination Versus Dorzolamide 1%/Timolol 0.5% in Patients With Open-Angle Glaucoma and Ocular Hypertension
Brief Title: Comparison of Intraocular Pressure (IOP)-Lowering Efficacy and Safety of AZORGA® Ophthalmic Suspension and COSOPT® Ophthalmic Solution
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Alcon, a Novartis Company (Industry)
Responsible Party: Sponsor
Organization: Alcon Research (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: ALJ-P2014-1; UMIN000017569 (Registry Identifier: UMIN)
Record Dates: First submitted 2014-12-22; First posted 2014-12-25 (Estimated); Results first posted 2016-12-08 (Estimated); Last update posted 2016-12-08 (Estimated); Status verified 2016-10

CONDITIONS: Open-Angle Glaucoma; Ocular Hypertension
Keywords: Open-angle glaucoma (OAG); Ocular hypertension (OHT); AZORGA®; COSOPT®
MeSH Terms: conditions — Glaucoma, Open-Angle; Ocular Hypertension | interventions — brinzolamide; Timolol; dorzolamide; Ophthalmic Solutions; dorzolamide-timolol combination

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- BRI/TIM (Experimental): Brinzolamide 1%/Timolol maleate 0.5% fixed combination ophthalmic suspension, 1 drop in each eye twice daily, and habitual PGA monotherapy, 1 drop in each eye once daily for 8 weeks.
  Interventions: Drug: Brinzolamide 1%/Timolol maleate 0.5% fixed combination ophthalmic suspension; Drug: Subject's habitual PGA monotherapy
- DOR/TIM (Active Comparator): Dorzolamide hydrochloride 1%/Timolol maleate 0.5% ophthalmic solution, 1 drop in each eye twice daily, and habitual PGA monotherapy, 1 drop in each eye once daily for 8 weeks.
  Interventions: Drug: Dorzolamide hydrochloride 1%/Timolol maleate 0.5% ophthalmic solution; Drug: Subject's habitual PGA monotherapy

INTERVENTIONS:
Drug: Brinzolamide 1%/Timolol maleate 0.5% fixed combination ophthalmic suspension
  Other Names: AZORGA®
  Arms: BRI/TIM
Drug: Dorzolamide hydrochloride 1%/Timolol maleate 0.5% ophthalmic solution
  Other Names: COSOPT®
  Arms: DOR/TIM
Drug: Subject's habitual PGA monotherapy

SUMMARY:
The purpose of this study is to evaluate AZORGA® Ophthalmic Suspension compared to COSOPT® Ophthalmic Solution for IOP-lowering efficacy in subjects with open-angle glaucoma or ocular hypertension.

DETAILED DESCRIPTION:
After the screening examination, subjects were enrolled in the study and moved into the observation period. During the observation period, prostaglandin-analog (PGA) monotherapy was applied. After the observation period of 4 weeks or more, the baseline examination was performed. Subjects were then randomized and moved into the treatment period.

ELIGIBILITY:
Inclusion Criteria:

* Understand the nature of the study and sign informed consent.
* Diagnosis of open angle glaucoma or ocular hypertension.
* Currently on PGA monotherapy or PGA + alpha-1/beta blocker or PGA + alpha-2 agonist at screening visit, and allowed to instill only PGA for 4 weeks until the baseline visit.
* Intraocular pressure (IOP) ≥ 15 mmHg (at least one same eye) at the baseline visit.
* Other protocol-specified inclusion criteria may apply.

Exclusion Criteria:

* History of bronchial asthma, bronchospasm, or serious chronic obstruction pulmonary disease.
* Uncontrolled heart failure, sinus bradycardia, A-V block (II, III grade), cardiogenic shock, right heart failure due to pulmonary hypertension or congestive heart failure.
* History of hypersensitivity to any of the excipients of the study medications.
* Severe renal function disorders, diabetic ketoacidosis and metabolic acidosis, uncontrolled diabetes, or hepatic disorders.
* Corneal disorder or history of chronic, recurrent or current severe inflammatory eye disease in either eye.
* History of ocular trauma in either eye within 6 months prior to the screening examination.
* Ocular infection or ocular inflammation in either eye.
* History of or current clinically significant or progressive retinal disease in either eye.
* Intraocular surgery in either eye within 6 months prior to the screening examination.
* Ocular laser surgery in either eye within 3 months prior to the screening examination.
* Any abnormality preventing reliable applanation tonometry of either eye.
* Best-corrected visual acuity (BCVA) worse than 0.2 score (decimal visual acuity) in either eye.
* Severe visual field loss in either eye.
* Use of prohibited medication, as specified in the protocol.
* Pregnant, lactating, or intending to become pregnant during the study period.
* Currently on therapy or have been on therapy with another investigational agent within 30 days prior to the screening examination.
* History of or current evidence of a severe illness or any other condition which would make the subject, in the opinion of the investigator, unsuitable for the study.
* Other protocol-specified exclusion criteria may apply.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 218 (Actual)
Dates: Start 2014-12; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical and Regulatory Affairs, Study Director — Alcon Japan, Ltd.
Locations (1):
- Contact Alcon Japan Ltd. for Trial Locations, Tokyo, Japan

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from 26 study sites in Japan.
Pre-assignment Details: Of the 218 enrolled, 6 subjects withdrew informed consent and 11 were exited as screen failures prior to randomization. This reporting group includes all randomized subjects (201).
Groups:
- BRI/TIM: Brinzolamide 1%/Timolol maleate 0.5% fixed combination ophthalmic suspension, 1 drop in each eye twice daily, and habitual prostaglandin-analog (PGA) monotherapy, 1 drop in each eye once daily for 8 weeks.
Period: Overall Study
Arm/Group | BRI/TIM | DOR/TIM
Started | 98 | 103
Safety Set | 98 | 103
Full Analysis Set (FAS) | 98 | 101
Per Protocol Set (PPS) | 92 | 97
Completed | 94 | 100
Not Completed | 4 | 3
Not completed — Adverse Event | 4 | 1
Not completed — Physician Decision | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Population: This analysis population includes all randomized subjects who received study medication and completed at least 1 scheduled on-therapy study visit (Full Analysis Set).
Groups:
- Total: Total of all reporting groups
Arm/Group | BRI/TIM | DOR/TIM | Total
Number analyzed (Participants) | 98 | 101 | 199
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.1 (11.8) | 64.4 (12.3) | 63.7 (12.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 52 | 53 | 105
  Male | 46 | 48 | 94

OUTCOME MEASURES:

1. Primary Outcome: Least Squares Mean Change From Baseline in Intraocular Pressure (IOP) at 11 AM
Description: IOP (fluid pressure inside the eye) was assessed using Goldmann applanation tonometry and measured in millimeters of mercury (mmHg). Data from 4 and 8 weeks at 11 AM were pooled, and a negative change indicates an improvement. One eye (target eye) was used for the analysis.
Time Frame: Baseline (Day 0), Week 4, Week 8 at 11 AM
Population: This analysis population includes all subjects who received study medication and met inclusion/exclusion criteria prior to randomization (Per Protocol Set).
Measure: Least Squares Mean (95% Confidence Interval); unit: mmHg
Arm/Group | BRI/TIM | DOR/TIM
Number analyzed (Participants) | 92 | 97
mmHg
  Baseline | 17.0 [16.6 to 17.3] | 17.0 [16.6 to 17.3]
  Mean change pooled over Week 4 and Week 8 | -3.3 [-3.6 to -2.9] | -3.4 [-3.7 to -3.0]

2. Secondary Outcome: Least Squares Mean Change From Baseline in IOP at 9 AM
Description: IOP (fluid pressure inside the eye) was assessed using Goldmann applanation tonometry and measured in millimeters of mercury (mmHg). Data from 4 and 8 weeks at 9 AM were pooled, and a negative change indicates an improvement. One eye (target eye) was used for the analysis.
Time Frame: Baseline (Day 0), Week 4, Week 8 at 9 AM
Population: Per Protocol Set (PPS)
Measure: Least Squares Mean (95% Confidence Interval); unit: mmHg
Arm/Group | BRI/TIM | DOR/TIM
Number analyzed (Participants) | 92 | 97
mmHg
  Baseline | 17.4 [17.1 to 17.8] | 17.3 [17.0 to 17.7]
  Change at Pool (Week 4, Week 8) | -3.3 [-3.6 to -2.9] | -2.9 [-3.2 to -2.5]

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) were collected from time of informed consent throughout the duration of a subject's participation in the study (up to 8 weeks). Ocular adverse events are presented for both study eye and non-study eye combined. AEs are reported as pretreatment and treatment-emergent. This analysis population includes all subjects who received study medication (Safety Analysis Set).
Description: An AE was defined as all medically undesirable or unintended diseases or symptoms that occur in subjects who receive study medication regardless of the causal relationship. Reports of AEs were obtained through solicited and spontaneous comments from the subjects and through observations by the Investigator as outlined in the study protocol.
Groups:
- Pretreatment: All subjects who consented to participate in the study prior to the initiation of study treatment
Arm/Group | Pretreatment | BRI/TIM | DOR/TIM
Serious Adverse Events (participants affected / at risk) | 1/218 | 1/98 | 0/103
Other Adverse Events (participants affected / at risk) | 0/218 | 21/98 | 16/103
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pretreatment (N=218) | BRI/TIM (N=98) | DOR/TIM (N=103)
Appendicitis (Infections and infestations) | 1 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Pretreatment (N=218) | BRI/TIM (N=98) | DOR/TIM (N=103)
Blurred vision (Eye disorders) | 0 | 20 | 9
Eye irritation (Eye disorders) | 0 | 2 | 10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor reserves the right of prior review of any publication or presentation of information related to the study.